CLINICAL TRIAL: NCT00522743
Title: Two Arms, Open, Controlled, Prospective, Intervention Study to Evaluate the Growth and Metabolic Response to Growth Hormone and Gonadotropin-releasing Hormone Agonist Treatment Versus Growth Hormone Alone in Boys Born SGA
Brief Title: Growth and Metabolic Response to GH and GnRHa Treatment Versus GH Alone in Boys Born SGA.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Prof. Moshe Phillip, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rmc073243ctil; SGA boys 3243
Record Dates: First submitted 2007-08-29; First posted 2007-08-30 (Estimated); Last update posted 2010-07-14 (Estimated); Status verified 2010-07

CONDITIONS: SGA and Growth
Keywords: SGA; GH; GnRHa; IGF-1
MeSH Terms: interventions — Growth Hormone; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): GH & GNRHa treatment
  Interventions: Drug: growth hormone and gonadotropin-releasing hormone agonist
- 2 (Active Comparator): GH treatment
  Interventions: Drug: growth hormone

INTERVENTIONS:
Drug: growth hormone and gonadotropin-releasing hormone agonist — GH & GNRHa treatment
  Arms: 1
Drug: growth hormone — GH treatment
  Arms: 2

SUMMARY:
A 2-arms randomized open prospective intervention study to determine the Growth and metabolic response to growth hormone and gonadotropin-releasing hormone agonist treatment versus growth hormone alone in boys born SGA.

All subjects will be treated with NorditropinSimplex at a dosage of 100mcg/kg/d.

At onset of puberty, subjects will be randomized into either combined treatment with GH and GnRHa or GH alone.

DETAILED DESCRIPTION:
A 2-arms randomized open prospective intervention study including 20 boys, in order to determine the effect of growth hormone (GH) and gonadotropin-releasing hormone agonist treatment versus growth hormone (GnRHa) alone on growth and metabolic response.

Objectives:

The primary objective is to investigate the effect of delaying the pubertal process by pubertal suppression on growth and final height of boys who were born SGA and treated with GH.

The secondary objectives are to determine the metabolic effect of the combined therapy of GH plus gonadotropin agonists to that of GH alone on the dietary intake, serum leptin, ghrelin, IGF-1, lipid and lipoprotein concentrations prior to and during treatment, and to assess the quality of life between the two groups.

Study population:

20 prepubertal boys.

Inclusion Criteria:

1. Ages 10-13
2. IUGR
3. Height of at least 2 standard deviations below the mean height for chronological age and sex according to the 2000 standards from the Centers for Disease Control and Prevention (CDC).
4. prepubertal(Tanner stage 1) at commencement of trail.
5. Peak GH above 10ng/ml in at least one provocative test for GH secretion.
6. Signed informed consent form.

Exclusion criteria:

1. Growth retardation associated with malignancy, severe chronic disease, genetic syndromes and endocrine disorders.
2. Diabetes.
3. Treatment with any medical product which may interfere with GH effects.

Trail design:

A prospective, randomized controlled study assessing the impact of two years of combined treatment with GH and GnRHa on height of boys with severe growth failure due to SGA with height >2.25 SDS , compared with GH alone.

All subjects will be treated with NorditropinSimplex at a dosage of 100mcg/kg/d. At onset of puberty (testicular volume greater than 4 ml in consecutive examinations) subjects will be randomized into either combined treatment with GH and GnRHa or GH alone.

Methods:

1. Urine test will be held every three months.
2. X-ray photograph for bone age determination will be taken at baseline and every year after.
3. Blood will be taken at baseline and every year after in order to evaluate the following parameters: Lipid and lipoprotein concentrations, ghrelin, leptin, glucose, insulin and HbA1c.
4. Blood will be taken on randomization visit and three months after in order to evaluated the following parameters: LH, FSH and Testosterone
5. Blood will be taken at baseline and every half a year after to evaluate levels of IGF-1.
6. For evaluation of the growth hormone response, additional blood tests will be preformed one month and three months after treatment with growth hormone.
7. On every blood and urine that will be taken, proteomic analysis will be held.
8. Before treatment with growth hormone, one year after treatment and in the end of the study quality of life questionnaire, appetite questionnaire and Psychological questionnaires will be filled.

The safety of growth hormone treatment will be assessed from:

1. Monitoring of adverse events.
2. Measurement of HbA1c.
3. Measurement of hematology, serum biochemistry and urinalysis laboratory variables.
4. Measurement of fasting glucose and insulin concentrations.
5. IGF-1
6. Physical examinations and measurements of vital signs height and body weight.
7. Measurement of bone age.

ELIGIBILITY:
Inclusion Criteria:

1. Boys
2. IUGR
3. Ages 10-13
4. height of at list 2.0 standard deviations below the mean height for chronological age and sex according to the 2000 standards from the Centers for Disease Control and Prevention (CDC)
5. Prepubertal (tanner stage 1) at commencement of trail
6. Peak GH above 10ng/ml in at least one provocative test for GH secretion 7.Signed informed consent

Exclusion Criteria:

1. Growth retardation associated with malignancy, severe chronic disease, genetic syndromes and endocrine disorders
2. Diabetes
3. Treatment with any medical product which may interfere with GH effects

Ages: 9 Years to 13 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2005-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Height measurements | every 3 monthes, during all study period

SECONDARY OUTCOMES:
IGF-1 concentration | every 6 monthes, during all study period
Hormone profile, Lipid and lipoprotein concentrations | once a year during all study period
Prepubertal changes | every 3 monthes during all study peiod
Bone age | once a year, during all study period
quality of life questionnaire | once a year, during all study period
Psychological questionnaire | once a year, during all study peiod

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Phillip, Professor, Principal Investigator — Rabin Medical Center
Locations (1):
- Schnider children medical center, Petah Tikva, Israel